CLINICAL TRIAL: NCT07302243
Title: Association Between One Lung Ventilation and Myocardial Injury Markers (Troponin T and I) in Thoracic Surgical Procedures : An Observational Cohort Study (OLVTIS)
Brief Title: Association Between One Lung Ventilation and Myocardial Injury Markers (Troponin T and I) in Thoracic Surgical Procedures (OLVTIS)
Acronym: OLVTIS
Status: Completed | Type: Observational
Sponsor: Universitas Jenderal Soedirman (Other)
Collaborators: RS Prof. Dr. Margono Soekardjo Purwokerto (Unknown)
Responsible Party: Principal Investigator, MM Rudi Prihatno, Consultant Neuroanesthesiologist and Dean, Faculty of Medicine, Jenderal Soedirman University, Universitas Jenderal Soedirman
Other Study IDs: UNSOED - OLV; 108/KEPK/PE/2025 (Other: Registry ID: The Research Ethics Commmite Faculty Medicine Jenderal Soedirman University)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Thoracic Anesthesia; One Lung Ventillation (OLV)
Keywords: one lung ventilation; thoracic surgery; troponin; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracotomy OLV: A single cohort of adult patients undergoing thoracotomy with one-lung ventilation. All participants receive standard general anesthesia. No interventions are assigned. Preoperative and postoperative cardiac biomarkers (Troponin T and I) and arterial blood gases are collected to evaluate myocardial injury associated with OLV.

SUMMARY:
This prospective single-group cohort study aims to investigate the association between the One-Lung Ventilation (OLV) technique and myocardial injury, as measured by postoperative Troponin T and Troponin I levels, in patients undergoing thoracic surgery. All eligible participants will undergo standardized anesthesia and OLV techniques, with cardiac biomarkers collected before surgery and six hours postoperatively. The findings of this study are expected to provide a better understanding of the impact of OLV on myocardial stress or injury during thoracic surgical procedures.

DETAILED DESCRIPTION:
The one-lung ventilation (OLV) technique offers significant operative advantages but may cause various physiological complications that can potentially affect cardiovascular function. Intraoperative hemodynamic changes may lead to postoperative myocardial infarction and increase mortality risk. Aim To determine the differences in postoperative troponin T and I levels in thoracic surgery with OLV. This cohort study involved thirty nine patients who underwent thoracic surgery with OLV. All subjects received OLV with a ventilation ratio of 50% air to 50% oxygen, a tidal volume of 5-6 mL/kg body weight, and a respiratory rate of 12 breaths per minute. Troponin T and I levels were measured before and after surgery. Hemodynamic status and perioperative parameters were recorded.

Here is a clear, structured English version suitable for the Study Description → Detailed Description section of ClinicalTrials.gov:

-

Detailed Study Procedures

Eligible participants who meet the study criteria will be identified by the research team. Each participant will receive a detailed explanation of the study objectives and procedures. Those who agree to participate will be asked to sign an informed consent form during the preoperative visit. all participants will undergo standard monitoring placement, including vital sign monitors and arterial line insertion. Patients will then be prepared for anesthesia induction.

Before the thoracic surgical procedure, baseline measurements will be obtained, including arterial blood gas (ABG) analysis and serum Troponin T and I levels.

All participants will receive general anesthesia. Induction will be performed using sufentanil (10-15 mcg), propofol (1.5-2.5 mg/kg), and rocuronium (0.6-1.2 mg/kg). Anesthesia maintenance will include sevoflurane (1-2%) and sufentanil infusion (5-20 mcg/hour). The anesthesia will be administered by anesthesia residents (5th semester or above) under supervision of an attending anesthesiologist.

Following successful endotracheal intubation using a double-lumen tube, mechanical ventilation will begin with a 50% oxygen and 50% air mixture. During two-lung ventilation, tidal volume will be set to 8 mL/kg with a respiratory rate of 12 breaths per minute. During one-lung ventilation (OLV), tidal volume will be adjusted to 5-6 mL/kg while maintaining a respiratory rate of 12 breaths per minute.

Throughout the surgical procedure, participants will undergo continuous hemodynamic monitoring. Additional intraoperative data, including duration of OLV and estimated blood loss, will be recorded. After surgery, patients will be transferred to the Intensive Care Unit (ICU) for postoperative monitoring.

All research participants will receive postoperative analgesia using a continuous sufentanil infusion at 0.1 mcg/kg/hour via syringe pump. Six hours after completion of the thoracic surgical procedure, postoperative ABG analysis and serum Troponin T and I levels will be obtained in the ICU. All collected research data will be documented, tabulated, and subsequently analyzed according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years who requiring surgical thoracotomy with one lung ventilation
* Classified as ASA Physical Status I - III
* Provide Informed concent ( patient or legal representative)

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Patients who refuse to participate in the study
  * Patients undergoing thoracotomy surgery involving manipulation of the cardiovascular system
  * Patients with a history of heart disease and/or current cardiac treatment
  * Patients with severe hepatic or renal impairment
  * Patients with contraindications or allergies to the medications used in the study
  * Pregnant or Lactating women
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Troponin T Levels Pre- and Post-Thoracotomy with One-Lung Ventilation | Pre operative baseline and 6 - 12 hours post operative
  Troponin T levels are measured before surgery and again 6-12 hours after the thoracotomy procedure to evaluate myocardial injury potentially associated with one-lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Adeastri Hapsari, M.D, Principal Investigator — Department of Anesthesiology and Intensive Care, Faculty of Medicine Jenderal Soedirman University / RSUD Prof. Dr. Margono Soekarjo Purwokerto. Purwokerto, Indonesia
Locations (1):
- RSUD Prof. Margono Soekarjo, Purwokerto, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared because of institutional privacy policy and ethical considerations involving patient data from RSUD Prof. Dr. Margono Soekarjo Purwokerto.